CLINICAL TRIAL: NCT01554878
Title: Observational Studies, Prospective, Multicenter, to Evaluate the Effect of Treatment of Knee Osteochondral Lesions of Outerbridge Grade III-IV
Brief Title: Observational Study on the Treatment of Knee Osteochondral Lesions of Grade III-IV
Acronym: LOGIC
Status: Completed | Type: Observational
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ESREFO08
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2014-05

CONDITIONS: Degenerative Lesion of Articular Cartilage of Knee
Keywords: osteochondral defect of the knee

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- knee surgery
  Interventions: Procedure: knee surgery

INTERVENTIONS:
Procedure: knee surgery — Reparative, replacement or regenerative techniques, with or without associated osteotomy.

SUMMARY:
The purpose of the study is to evaluate prospectively the outcome of treatment interventions of knee osteochondral lesions Outerbridge grade III and IV.

DETAILED DESCRIPTION:
The main purpose of the study is to prospectively evaluate the outcome of treatment interventions with replacement, repair and regenerative approaches, of osteochondral articular lesions or defects, Outerbridge grade III and IV, in terms of symptomatic and functional recovery 12 months after surgery.

ELIGIBILITY:
Inclusion criteria:

patients referred to the participating centers for symptomatic treatment of degenerative lesions of the knee, which meet the following inclusion criteria:

* symptomatic osteochondral lesions of grade III or IV (according to classification of Outerbridge;
* Axial deviation with chondral damage, correct or not;
* Consent to the processing of personal data, signed and dated by patient;
* Patients of both sexes and aged between 30 and 60 years;
* Patients willing to participate actively in the rehabilitation program and to attend post-operative follow-up visits.

Exclusion criteria:

* Patients with synovitis;
* BMI> 30;
* Allergy to collagen or calcium phosphate;
* Patients with neoplastic disease;
* Patients with metabolic disorders, thyroid diseases, immune system disorders.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients referred to the participating centers for the treatment of symptomatic degenerative lesions of the knee, which meet the following inclusion criteria
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Score | 12 months post procedure
  Primary outcome measure will be the outcome of innovative treatments with repairing, regenerative and replacement techniques, with or without associated osteotomy, of knee osteochondral severe lesions(Outerbridge grade III and IV) in terms of symptoms improvement as assessed by means of the International Knee Documentation Committee (IKDC) subjective Knee Evaluation Score at 12 months postoperatively.

SECONDARY OUTCOMES:
functional recovery at International Knee Documentation Committee(IKDC) knee Examination | 12 months
Physical performance at Tegner activity score | 12 months post surgery
functional activity on the Lysholm Knee Scale | 12 months post surgery
Tissue regeneration at magnetic resonance (MRI) | 12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Raul Zini, MD, Study Director — Maria Cecilia Hospital; Luisangelo Sordo, MD, Principal Investigator — MARIA PIA HOSPITAL; Maurizio Bellettato, MD, Principal Investigator — SAN PIER DAMIANO; Andrea Mocci, MD, Principal Investigator — ANTHEA HOSPITAL
Locations (4):
- Italy (4):
  - Andrea Mocci, Bari, Bari
  - Raul Zini, Cotignola, Ravenna
  - Maurizio Bellettato, Faenza, Ravenna
  - Luisangelo Sordo, Torino, Torino

IPD SHARING:
Plan to Share IPD: No